CLINICAL TRIAL: NCT04341558
Title: Family SuppleMented pAtient monitoRing afTEr suRgery: A Pilot Trial
Acronym: SMARTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Busitema University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: QMERC2019/72
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-02

CONDITIONS: Postoperative Care; Vital Signs

STUDY DESIGN:
Intervention Model Description: Single-centre stepped-wedge cluster randomised trial conducted in four surgical wards over a six-month period
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline (No Intervention): During this baseline period, postoperative monitoring will be continued as normal by nursing and medical staff without intervention. No training of family members will take place
- Intervention (Active Comparator): Family carers will be trained to perform and document basic vital signs whilst they provide personal care to their relatives after surgery in order to supplement patient monitoring conducted by nursing staff.
  Interventions: Other: Family supplemented patient monitoring

INTERVENTIONS:
Other: Family supplemented patient monitoring — Intervention training sessions will last 30 minutes and will be held twice a day over a period of six months. Carers will be welcome to attend as often as they wish. Carers will be given practical training to assess the following vital signs: heart rate, respiratory rate, conscious level (AVPU scale) and arterial oxygen saturation (SpO2) in accordance with trial standard operating procedures. An important component of the training package will be ensuring carers know how to wash their hands before and after contact with their patients. The study team will ensure that handwashing facilities are available on the ward for use by carers. Carers will record vital signs on a basic observation chart every 4 hours after surgery. They will compare results with colour posters displayed throughout each ward, providing guidance on how and when to notify nursing staff of abnormal vital signs.
  Arms: Intervention

SUMMARY:
To develop an intervention to train family carers to perform and document basic vital signs whilst they provide personal care to their relatives after surgery in order to supplement patient monitoring conducted by nursing staff. To evaluate the effect of this intervention on the frequency of documented vital signs for patients in the first three days after surgery in a stepped-wedge cluster trial.

DETAILED DESCRIPTION:
Quality improvement (QI) interventions can be seen has having a 'hard core', the clinical processes or practices that are the focus of improvement, and a 'soft periphery', the improvement methods that will enable change to occur. In the SMARTER trial, family carers will be trained to perform basic vital signs monitoring and document the results. Nursing and medical teams looking after patients on the wards will retain full responsibility for patient care throughout all phases of the trial. The nursing team will be provided with an identical observation chart for all their ward patients at the beginning of the trial and will be given training on how to use them and how to respond to deteriorating vital signs.

During the intervention period, in addition to the nurses' vital signs monitoring, family members will be asked to perform basic vital signs monitoring. Participants will be given clear guidance on when to alert staff to potential danger signs.

The soft periphery is the training programme and resources designed to assist staff to rapidly and effectively train these skills combined with ongoing maintenance strategies to ensure the compliance with the intervention is maintained throughout the intervention period. The investigators will use the Medical Research Council (MRC) Complex Intervention framework to guide the development and evaluation of our intervention. Previous empirical work on task-sharing and relevant theory will be used to design the intervention and associated programme theory (Phase 1 of the MRC framework), with an iterative co-design process used to further develop these and test how the intervention works in practice (Phase 2).

Intervention training sessions will last 30 minutes and will be held twice a day over a period of six months. Participants will be welcome to attend as often as they wish. Participants will be given practical training to assess the following vital signs: heart rate, respiratory rate, conscious level (AVPU scale) and arterial oxygen saturation (SpO2) in accordance with trial standard operating procedures. An important component of the training package will be ensuring participants know how to wash their hands before and after contact with their patients. The investigators will ensure that handwashing facilities are available on the ward for use by participants. Participants will record vital signs on a basic observation chart every 4 hours after surgery. They will compare results with colour posters displayed throughout each ward, providing guidance on how and when to notify nursing staff of abnormal vital signs.

Participants will have access to the following equipment throughout the trial: pulse oximeter, wall clock, colour coded guidelines on wall, observation charts, clipboard and pen. Although poor numeracy and literacy are common in eastern Uganda, most patients will have a carer who is able to read a digital clock and write numbers. The observation chart will be designed to be very simple to use. Participants will be encouraged to attend the training sessions each day to ensure their skills and knowledge are refreshed. After the third post-operative day, the trial intervention will end although participants may choose to continue monitoring vital signs and attending training sessions if they wish. It is acknowledged that carers may have to change throughout the day due to conflicting family or work commitments. Participants will be encouraged to remain available to monitor their patients for the duration of the study period (72 hours). Medical and nursing staff on the wards will undergo training in how to respond appropriately to abnormal vital signs.

ELIGIBILITY:
Inclusion Criteria:

Patients:

• Patients ≥5 years of age undergoing surgery at Mbale Regional Referral Hospital, who receive post-operative care in one of four main surgical wards, with a family carer prepared to participate in the trial intervention.

Carers:

* All carers will be included in the trial if they feel they are capable of performing and documenting the basic vital signs provided they agree to participate in the trial.
* The ability to speak English, Luganda, Lugisu, Ateso or Lugwere
* The ability to read a digital clock (to measure vital signs)
* Numeracy sufficient to write numbers on the basic observation chart

Exclusion Criteria:

Patients:

* Refusal of informed consent.
* Identification of potential participant >24hours after operative procedure has taken place

Carers:

• Refusal of informed consent.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1395 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Frequency of documented vital signs for patients after surgery | 72 hours
  To develop a training and support intervention, in accordance with the MRC complex intervention framework, to train family carers to perform and document basic vital signs, to supplement routine monitoring of patients by nursing staff, whilst they provide personal care to their relatives after surgery and to evaluate the effect of this intervention on frequency of documented vital signs for patients in the first three days after surgery in a stepped-wedge cluster trial (explanatory outcome).

SECONDARY OUTCOMES:
Duration of hospital stay | 30 days
  To evaluate the impact of the intervention on the duration of patients' length of hospital stay
All cause mortality at 30 days | 30 days
  To evaluate the effect of the intervention on in-patient mortality, to inform the design of a subsequent international clinical trial across Africa

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Pearse, MD, Principal Investigator — Queen Mary University of London
Locations (1):
- Mbale Regional Referral Hospital, Mbale, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hewitt-Smith A, Bulamba F, Patel A, Nanimambi J, Adong LR, Emacu B, Kabaleta M, Khanyalano J, Maiga AH, Mugume C, Nakibuule J, Nandyose L, Sejja M, Weere W, Stephens T, Pearse RM. Family supplemented patient monitoring after surgery (SMARTER): a pilot stepped-wedge cluster-randomised trial. Br J Anaesth. 2024 Oct;133(4):846-852. doi: 10.1016/j.bja.2024.06.027. Epub 2024 Jul 27. PMID 39069451